CLINICAL TRIAL: NCT06109961
Title: Hyperbaric Oxygen Therapy for Perianal Fistulizing Crohn's Disease Not Responsive or Intolerant to Conventional Care: HYPNOTIC Pilot Study
Acronym: HYPNOTIC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRRF ID 5207
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: Perianal Crohn's disease (PCD); Hyperbaric oxygen therapy (HBOT); Tumor necrosis factor (TNF)
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Oxygen; Standard of Care

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, randomized open-label clinical trial and parallel registry.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Hyperbaric Oxygen Therapy (Experimental): The active Hyperbaric Oxygen Therapy (HBOT) arm will receive 100% oxygen at 2.0-2.5 atmospheres (ATM).
  Interventions: Drug: Oxygen Gas for Inhalation
- Standard of care treatment (Other): The standard of care for perianal Crohn's disease (PCD) involves conventional therapies such as immunosuppressive agents and biologics, which can be used to induce and maintain fistula remission. Tumor necrosis factor (TNF) antagonists are considered the first-line therapy for PCD, and clinical trial evidence supports their efficacy in achieving short-term fistula remission.
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Oxygen Gas for Inhalation — The active Hyperbaric Oxygen Therapy (HBOT) arm will receive 100% oxygen at 2.0-2.5 atmospheres (ATM).
  Arms: Active Hyperbaric Oxygen Therapy
Other: Standard of care — The accepted standard of care for perianal Crohn's disease (PCD) involves conventional therapies such as immunosuppressive agents and biologics, which can be used to induce and maintain fistula remission.
  Other Names: Conventional therapies
  Arms: Standard of care treatment

SUMMARY:
This study aims to test a new treatment called hyperbaric oxygen therapy (HBOT) for a severe type of inflammatory bowel disease called perianal Crohn's disease (PCD). PCD causes painful perianal infections and chronic drainage from fistula tracts, and current treatments are only moderately effective and may not be suitable for all patients. HBOT is a safe and commonly used treatment for chronic non-healing wounds and other conditions. Previous studies have suggested that HBOT may help heal fistulas in PCD patients, but these studies were small and lacked controls.

DETAILED DESCRIPTION:
Hyperbaric oxygen therapy (HBOT) is an effective intervention for improving healing of chronic wounds. HBOT involves the delivery of 100% oxygen in a pressurized environment, typically two to three times standard atmospheric pressure at sea level (2.0-2.5 ATA). This results in increased oxygen tension in plasma and promotes the diffusion of oxygen into tissue, which stimulates tissue restorative pathways that are essential for wound healing16. Hyperoxia also modulates the immune system by suppressing proinflammatory cytokines and promoting the production of anti-inflammatory cytokines. It also enhances the production of growth factors, mobilize stem cells, and stimulates anti-microbial pathways, all of which are believed to be central mechanisms involved in the repair of damaged tissue in IBD. The safety profile of HBOT is also excellent, with a reported adverse event incidence of 10 per 10,000. The most reported adverse event is middle ear barotrauma, which is minor and not life threatening.

There is emerging evidence that HBOT may be an effective treatment option for perianal Crohn's disease (PCD). To date, 10 observational studies with a total of 118 patients with PCD refractory to conventional therapy have assessed the effectiveness and safety of HBOT (McCurdy et al., IBDJ 2021). In this small number of patients, HBOT resulted in high rates of clinical response (75% [95% CI, 66%-83%; I2, 0]) and clinical remission (55% [95% CI, 44%-65%; I2, 61]) (Figure 1). Additionally, the HOT-TOPICs study, an open-label observational study demonstrated that HBOT was associated with radiologic improvement of fistula tracts as shown by a reduction in the modified Van Assche MRI score from 9.2 (95% CI, 7.3-11.2) to 7.3 (95% CI, 6.9-9.7). Despite these encouraging results, formal controlled clinical trials have not yet been conducted in patients with PCD to determine the true clinical impact of HBOT in this disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>17 years old)
* Diagnosis of Crohn's disease based on standard endoscopic, radiologic and/or histologic criteria.
* One or more perianal fistula tract connecting the rectum and the perianal skin. Patients must have active fistula drainage and/or a recurrent perianal abscess within the past month.
* Failure or intolerance of conventional therapy (imuran, methotrexate, anti-TNF therapies, vedolizumab and/or ustekinumab). Failure is defined as persistent perianal drainage or recurrent abscesses after a minimum of 3 months of therapy.
* Standard or care treatment has been stable (dose and treatment interval) for at least 3 months.
* Able to provide written consent to participate

Exclusion Criteria:

* Fistulas not believed to be due to Crohn's disease (examples include, obstetrical complications, tuberculosis, anorectal cancer or diverticular fistula).
* Rectovaginal fistulas.
* Undrained perianal abscesses on pelvic MRI exams (abscesses will require successful drainage by an exam under anaesthesia with or without seton prior to study inclusion).
* Surgical procedure such as an advancement flap, fistula plug, fistula glue or ligation of intersphincteric fistula tract (LIFT) procedure within the past 6 months.
* Diverting ostomies or ileal pouch anal anastomosis.
* Current or planned pregnancy or lactation during the study treatment period.
* Contraindications to HBOT (claustrophobia, incompatible implanted medical device, and other conditions) based on the discretion of our HBOT clinicians.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1 recruitment rate | 1 year
  Primary outcome for phase 1 is the rate of recruitment. Recruitment is defined as the number of randomized patients that receive at least one treatment (active HBOT or control) per year. After one year, recruitment of 20 patients or more (an average of 4 patients per site) will be considered acceptable to proceed to phase 2 without a requirement for modifications, recruitment of 10-20 patients will suggest minor modifications to the protocol are required and recruitment of less than 10 patients will suggest major modifications to the protocol are required prior to proceeding to phase 2.

SECONDARY OUTCOMES:
Phase 2 numbers of closure all external openings of fistula tracts | 1 year
  The primary outcome for phase 2 is the proportion of patients who achieve combined remission of perianal fistulizing Crohn's Disease at week 12 defined as closure of all external openings by finger compression test, and an absence of collections >2 cm confirmed by MRI assessment assessed at 8-12 weeks. MRI pelvis is the optimal outcome measure for measuring response to treatment as it has been shown to be the most accurate test for predicting long-term outcomes.